CLINICAL TRIAL: NCT00657826
Title: ATS 3f(r) Aortic Bioprosthesis Model 1000
Brief Title: ATS 3f(r) Aortic Bioprosthesis Model 1000, 19mm
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision to end study due to limited enrollment and study population
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001 Rev. E
Record Dates: First submitted 2008-04-04; First posted 2008-04-14 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Heart Valve Diseases
Keywords: Diseased Heart Valve, Replacement
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 19mm arotic valve implant (Experimental): Single arm study for patients who require a smaller valve size of the ATS 3f® Aortic Bioprosthesis, Model 1000, 19mm.
  Interventions: Device: ATS 3f® Aortic Bioprosthesis, Model 1000, 19mm

INTERVENTIONS:
Device: ATS 3f® Aortic Bioprosthesis, Model 1000, 19mm — Isolated aortic valve replacement with a size 19mm valve

SUMMARY:
The initial clinical investigation titled "ATS 3f(r) Aortic Bioprosthesis Model 1000 Study," was a prospective, non-randomized, multi-center study designed to evaluate the the safety and effectiveness obtained from 800 patient years using a common clinical protocol. Twenty-three (23) sites internationally and in the United States combined enrolled 405 patients. The objective of the study was to evaluate the safety and effectiveness of the ATS 3f(r) Aortic Bioprosthesis Model 1000 equine pericardial prosthesis in a a patient population undergoing isolated aortic valve replacement of his / her native aortic valve, or replacement of a failed prosthesis with or without concomitant procedures.

Addendum: After receiving PMA approval in October of 2008 of the 21mm-29mm sizes, this IDE was expanded to comply with the conditions set forth in the approval notice. Study Protocol S2001 Rev. E is a continuation of the original protocol, but is only enrolling subjects who require a 19mm ATS 3f(r) Aortic Bioprosthesis, Model 1000 and is described as "A multi-center, non-randomized trial, designed to obtain 800 patient years. Each enrolled patient will be followed for a minimum one year and annually thereafter until size 19mm product approval or study cessation. Preoperative, discharge or 30 days (which ever comes last), 3-6 month, and annual follow-up data are required.

DETAILED DESCRIPTION:
The patients for whom ATS Medical, Inc., ATS 3f(r) Aortic Bioprosthesis Model 1000 is intended are those patients whose prognosis without surgery for replacement of the diseased natural valve or previous implanted prosthetic valve is unacceptably poor in terms of survival, quality of life, or both, in the opinion of the attending physicians. For this special subset of patients, there are a number of widely accepted prosthetic heart valves in use.

ELIGIBILITY:
Inclusion Criteria:

* This patient requires isolated aortic valve replacement with or without concomitant procedures such as coronary artery bypass or another valve reconstruction. (The three remaining valves must be of native tissue).
* This patient is sufficiently ill to warrant replacement of his/her diseased natural or prosthetic valve, based on standard cardiovascular diagnostic workups.
* This patient is in satisfactory condition, based on the physical exam and investigator's experience, to be an average or better operative risk, (i.e., likely to survive one year postoperatively).
* This patient is geographically stable and willing to return to the implant center for follow-up visits.
* This patient has been adequately informed and consents to his/her participation in the clinical study, and of what will be required of him/her, in order to comply with the protocol.

Exclusion Criteria:

* This patient is twenty (20) or less than twenty years of age.
* This patient has a non-cardiac major or progressive disease, which in the investigator's experience produces an unacceptable increased risk to the patient, or results in a life expectancy of less than 12 months.
* This patient is an intravenous drug and/or alcohol abuser.
* This female patient is pregnant (urine HCG test result positive), or lactating.
* This patient presents with active endocarditis.
* This patient presents with congenital bicuspid aortic anatomy.
* This patient has a previously implanted prosthetic valve that is not being replaced by a study valve.
* This patient requires mitral, tricuspid or pulmonic valve replacement.
* This patient is participating in concomitant research studies of investigational products.
* This patient will not agree to return to the implant center for the required number of follow-up visits or is geographically unavailable for follow-up.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2001-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
NYHA Functional Classification | 3-6 months, 11-14 months, anuually for a minimum of 800 patient years to support a PMA application to the U.S. FDA
  The NYHA classifications will be analyzed to demonstrate if implanting of the study valve leads to an improvement in this clinical parameter for the patient.
Blood Data | 3-6 months, 11-14 months, anuually for a minimum of 800 patient years to support a PMA application to the U.S. FDA
  Blood data will be analyzed preoperatively and postoperatively to deomonstrate if implanting of the study valve results in acceptable parameters for SLDH, Haptoglobin, Hematocrit and Reticulocyte parameters. Platelet and white blood cell count will also be analyzed.
Cardiovascular Complications | 3-6 months, 11-14 months, anuually for a minimum of 800 patient years to support a PMA application to the U.S. FDA
  All cardiovascular related complications should be conducted and evaluated according to the STS guidelines. In reporting complications, all cardiovascular related symptoms will be evaluated as to their relation to the valve.
Hemodynamic Performance | 3-6 months, 11-14 months, anuually for a minimum of 800 patient years to support a PMA application to the U.S. FDA
  Assessment of hemodynamic performance shall include analysis of Doppler echocardiographic studies at the early and late postoperative evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Palmer, Study Director — Medtronic
Locations (2):
- Lankenau Institute for Medical Research, Wynnewood, Pennsylvania, United States
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Medtronic, Inc. Corporate website — http://www.medtronic.com/